CLINICAL TRIAL: NCT01661582
Title: Myocardial Ischaemia After Exposure to Diesel Exhaust
Acronym: MIDAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: National Institute for Public Health and the Environment (RIVM) (Other Government); British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MIDAS
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Coronary Heart Disease
Keywords: Air Pollution; Myocardial Ischaemia; Coronary Blood Flow; Diesel Exhaust; Troponin; Electrocardiography
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Filtered Air Exposure (Placebo Comparator): Subjects will be exposed to filtered air for 1 hour during intermittent exercise in a purpose-built exposure facility
  Interventions: Other: CT/PET Myocardial Perfusion Imaging using O-15 water; Other: Coronary blood flow measured by doppler echocardiography
- Dilute Diesel Exhaust Exposure (Experimental): Subjects will be exposed to dilute diesel exhaust (~300 mcg/m3) for 1 hour during intermittent exercise in a purpose-built exposure facility
  Interventions: Other: CT/PET Myocardial Perfusion Imaging using O-15 water; Other: Coronary blood flow measured by doppler echocardiography

INTERVENTIONS:
Other: CT/PET Myocardial Perfusion Imaging using O-15 water
Other: Coronary blood flow measured by doppler echocardiography

SUMMARY:
Exposure to particulate air pollution is associated with increases in cardiovascular mortality and morbidity. The pathophysiological mechanisms underlying this observation are emerging, and exposure to particulate air pollution has been shown to result in increases in blood pressure and arterial tone, impaired vascular function and an increased tendency for blood to clot as well as an increase in atherosclerotic plaque burden. Recent evidence from panel studies and controlled exposure studies have suggested an increase in myocardial ischaemia (a reduction in blood flow to the heart) following exposure. In this study we aim to investigate directly myocardial (heart) blood flow following exposure to diesel exhaust (as a model of urban air pollution) using CT/PET myocardial perfusion imaging in male patients with stable coronary disease and healthy male controls. We hypothesize that following exposure to dilute diesel exhaust:

1. Myocardial blood flow will be reduced
2. Coronary flow reserve will be impaired
3. The magnitude of impairment will be higher in patients with coronary disease as compared to healthy controls

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers will be taking no regular medication, have a normal electrocardiogram and exercise stress test
* Patients with a previous history of myocardial infarction or successful coronary revascularization (PTCA or coronary artery bypass grafting) but without symptoms of angina pectoris will be recruited

Exclusion Criteria:

* Healthy volunteers:
* Regular medication
* Abnormal 12-lead electrocardiogram
* Abnormal exercise stress test
* Patients with coronary disease
* Acute coronary syndrome within past 3 months
* Impaired left ventricular function
* Significant valvular heart disease
* Left ventricular hypertrophy
* Resting conduction defect
* Digoxin use
* Renal impairment (eGFR <60 mL/min)
* Hepatic impairment
* Asthma

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-09-20 (Actual); Primary Completion 2015-02-13 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
Myocardial blood flow and coronary flow reserve measured by CT/PET O-15 imaging | Immediately following exposure
  Myocardial blood flow will be measured at rest and at peak adenosine stress using CT/PET O-15 myocardial perfusion imaging immediately following exposure to diesel exhaust and filtered air

SECONDARY OUTCOMES:
Coronary flow reserve determined using doppler echocardiography | 1 hour following exposure
  Coronary blood flow will be determined in the left anterior descending coronary artery using doppler echocardiography at rest and at peak adenosine stress 1 hour following exposure to diesel exhaust and filtered air
Ultra-sensitive cardiac troponin-I | Before, 2 and 24 hours following exposure
  Blood samples will be obtained for measurement of cardiac troponin-I
ST segment deviation on continuous 12-lead electrocardiography | During and for the 24 hours aftet exposure
  A 12-lead electrocardiogram will be continuously recorded using Holter ECG monitor

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, PhD FRCP, Study Chair — University of Edinburgh; Jeremy P Langrish, MB BCh MRCP, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh / NHS Lothian, Edinburgh, United Kingdom

REFERENCES:
- [Background] Mills NL, Tornqvist H, Gonzalez MC, Vink E, Robinson SD, Soderberg S, Boon NA, Donaldson K, Sandstrom T, Blomberg A, Newby DE. Ischemic and thrombotic effects of dilute diesel-exhaust inhalation in men with coronary heart disease. N Engl J Med. 2007 Sep 13;357(11):1075-82. doi: 10.1056/NEJMoa066314. PMID 17855668
- [Derived] Langrish JP, Watts SJ, Hunter AJ, Shah AS, Bosson JA, Unosson J, Barath S, Lundback M, Cassee FR, Donaldson K, Sandstrom T, Blomberg A, Newby DE, Mills NL. Controlled exposures to air pollutants and risk of cardiac arrhythmia. Environ Health Perspect. 2014 Jul;122(7):747-53. doi: 10.1289/ehp.1307337. Epub 2014 Mar 25. PMID 24667535